CLINICAL TRIAL: NCT04169568
Title: Non-invasive Blood Pressuring Monitoring in Patients With Osteogenesis Imperfecta: Does Circumferential Cuff Pressure Result in Fractures?
Brief Title: Osteogenesis Imperfecta Blood Pressure Study
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Alicia McCarthy, Nurse Practitioner, Nemours Children's Clinic
Other Study IDs: 1465218-3
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OI manual cuff BP: Patients with diagnosis of Osteogenesis Imperfecta from ages 1 to 35 who are admitted to our institution to the inpatient, non-ICU setting, following orthopedic surgery for spine surgery, upper or lower extremity realignment and IM rodding
  Interventions: Procedure: Manual cuff blood pressure

INTERVENTIONS:
Procedure: Manual cuff blood pressure — Blood pressure will be obtained using a sphygmomanometer. Only Registered Nurses will apply BP cuff after careful inspection of the upper extremity for bruising, swelling or tenderness.

SUMMARY:
Osteogenesis Imperfecta (OI) is a genetic disorder caused by mutations to the alpha-1 or alpha-2 chain of type I collagen. Clinically, the disorder is characterized by bones that fracture easily, often from little or no apparent trauma. There is no information about Some institutions perform blood pressure monitoring on these patients with a cuff, while other institutions avoid this method due to concern for fracture. Instead, they use alternative forms of monitoring such as an arterial line. These methods come with their own risks, including clotting, decreased perfusion, and pain. In addition, arterial lines require intensive (and more expensive) monitoring in a pediatric intensive care unit due to risk of dislodgement and rapid blood loss. These blood pressure monitoring recommendations for patients with OI do not appear to be based on strong evidence. Anecdotally, some patients and healthcare professionals report hearing about individuals with OI who have suffered fractures from blood pressure cuffs. However, this is not well documented in the medical literature. Regular and accurate blood pressure monitoring is particularly important in the postoperative period, due to blood loss and fluid shifts, as well as utilization of advanced pain management techniques that can potentially impact blood pressure.

DETAILED DESCRIPTION:
Introduction Osteogenesis Imperfecta (OI) is a genetic disorder caused by mutations to the alpha-1 or alpha-2 chain of type I collagen. There are eight forms of OI, ranging from type I through VIII, however in types V to VIII the symptoms and severity fall within the range of the first four types. Clinically, the disorder is characterized by bones that fracture easily, often from little or no apparent trauma. These patients require special care and handling to minimize risk of fracture, and often undergo multiple surgeries to stabilize fractures and prevent or correct bone deformities. However, specific guidelines and restrictions for care, including clinical and postoperative care, vary between patients and among institutions. Some institutions perform blood pressure monitoring with a circumferential cuff, while other institutions avoid this method due to concern for iatrogenic fracture. Instead, they utilize alternative forms of monitoring such as an arterial line. Currently at Nemours, children and adults with OI have arterial lines placed in the OR for the purpose of BP monitoring. These more invasive methods come with their own risks, including thrombosis, decreased perfusion, and pain. In addition, arterial lines require intensive (and more expensive) monitoring in a pediatric intensive care unit due to risk of dislodgement and rapid blood loss. These blood pressure monitoring recommendations for patients with OI do not appear to be based on strong evidence. Anecdotally, some patients and healthcare professionals report hearing about individuals with OI who have suffered fractures from blood pressure cuffs. However, this is not well supported in the literature. Regular and accurate blood pressure monitoring is particularly important in the postoperative period, due to blood loss and fluid shifts, as well as utilization of advanced pain management techniques that can potentially impact blood pressure.

Aim of the study: In this observational study, we intend to evaluate the feasibility of non-invasive cuff blood pressure monitoring in a select group of patients with OI in the inpatient postoperative period.

Materials and Methods Following Nemours IRB approval and consent from the parent or legal guardian, fifty children with OI scheduled for lower extremity surgery with subsequent in-hospital admission will be enrolled in the study. Since we performed preformed lower extremity surgeries on thirty patients in each of the past two years, we anticipate the study will take two years to complete.

A group of registered nurses would be educated about the study and equipment used, review of appropriate blood pressure cuff size selection, blood pressure monitoring protocol, signs and symptoms of adverse events, and steps to take if an adverse event occurred.

Inclusion Criteria:

* Patients with OI who are undergoing extremity surgery or spinal fusion surgery.
* Patients between the ages of 1 and 35 years with OI who are admitted at our institution to a non-ICU inpatient setting in the postoperative period following an orthopedic surgery.
* Patients who initially require ICU-level care but transition to a non-ICU setting following an orthopedic surgery.
* Recent fracture in contralateral upper extremity (< 8 weeks, or upper extremity fracture that is not yet completely healed).
* Must be able to tolerate upper extremity blood pressures.
* Medical clearance by OI physicians (Kruse, Franzone) after review of fracture history, surgical procedures, x-rays.

Exclusion Criteria:

* Parent or child refusal, uncooperative child.
* History of frequent upper extremity fracture on ipsilateral side, or recent upper extremity fracture on ipsilateral side if only that side may be used.
* Clinical presence of thrombocytopenia (excessive or easy bleeding or bruising), admission or transfer to PICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients with OI who are undergoing extremity surgery or spinal fusion surgery.
* Patients between the ages of 1 and 35 years with OI who are admitted at our institution to a non-ICU inpatient setting in the postoperative period following an orthopedic surgery.
* Patients who initially require ICU-level care but transition to a non-ICU setting following an orthopedic surgery.
* Recent fracture in contralateral upper extremity (< 8 weeks, or upper extremity fracture that is not yet completely healed).
* Must be able to tolerate upper extremity blood pressures.
* Medical clearance by OI physicians (Kruse, Franzone) after review of fracture history, surgical procedures, x-rays.

Exclusion Criteria:

* Parent or child refusal, uncooperative child.
* History of frequent upper extremity fracture on ipsilateral side, or recent upper extremity fracture on ipsilateral side if only that side may be used.
* Clinical presence of thrombocytopenia (excessive or easy bleeding or bruising), admission or transfer to PICU.

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients between the ages of 1 and 35 with a diagnosis of Osteogenesis Imperfecta.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
Sphygmomanometer blood pressures | Every 4 hours for first 24 hours, then every 8 hours until discharge
  Cuff blood pressure measurements obtained without injury to patient with Osteogenesis Imperfecta

CONTACTS AND LOCATIONS:
Overall Officials: Alicia McCarthy, MSN, Principal Investigator — Nemours Children's Hospital
Locations (1):
- Nemours / A I duPont Hospital for Children, Wilmington, Delaware, United States